CLINICAL TRIAL: NCT06404502
Title: Feasibility and Acceptability of PRISMA for Prisoners in Switzerland - a Pilot Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of PRISMA for Prisoners in Switzerland
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-Nr. 2023-01378-pilot
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Psychological Distress; Anxiety; Depression; Suicidal Ideation
MeSH Terms: conditions — Anxiety Disorders; Depression; Suicidal Ideation | interventions — mesoglycan

STUDY DESIGN:
Intervention Model Description: The pilot RCT will inform us about the feasibility of PRISMA under usual practice conditions.
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions will be administered online.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISMA (Experimental): The intervention, PRISMA, addresses the issue of poor mental health of inmates during pretrial detention and after release. PRISMA has been adapted for the context of the model trial from Problem Management Plus (PM+). PRISMA has a total of four sessions provided during the first two weeks after entry such that most inmates can benefit from it before their potential release. The four sessions involve stress management, problem solving, meaningful activities (behavioral activation, and strengthening social support) and relapse prevention (staying well, looking forward). Additionally, participants will receive 2 booster sessions, 4 and 9 weeks after the final session.
  Interventions: Behavioral: PRISMA
- Control group (No Intervention): REGULAR PRETRIAL: participants in this group experience the same pretrial system, conditions, and services that they would have experienced if the RCT did not exist. They will not be offered PRISMA.

INTERVENTIONS:
Behavioral: PRISMA — PRISMA has been developed adapting PM+, a brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The adapted manual was developed to tailor the sessions to the structure of the Swiss prison system and the needs of inmates of jails in Switzerland. PRISMA involves the following elements: stress management, problem-solving, meaningful activities and relapse prevention
  PRISMA has four core features:
  * Evidence-based problem-solving strategies
  * Brief and easy to learn
  * Delivered by lay-helpers ("trainers")
  * Transdiagnostic, addressing depression, anxiety, stress, and practical problems as defined by participants;
  PRISMA has four sessions.
  Arms: PRISMA

SUMMARY:
In response to the significant mental health challenges faced by pretrial detainees, the Swiss Federal Justice Department has initiated a model trial in pretrial detention centres in Zurich and Bern. This model trial, named in German as a "Modellversuch," is designed to enhance detainees' wellbeing and evaluates various interventions through a randomized controlled trial. The "Prison Stress Management" (PRISMA) programme, a key intervention derived from the WHO's cognitive-behavioral therapy strategies, seeks to address the lack of mental health support within jails.

The goal of this pilot RCT is to evaluate the feasibility and acceptability of PRISMA for inmates inform a full-scale, definitive randomized controlled trial.

DETAILED DESCRIPTION:
Given the high prevalence of mental health issues, such as anxiety and depression, in pretrial detainees, the Swiss Federal Justice Department (SFJD) approved a model trial (in German named "Modellversuch Untersuchungshaft", MV). The MV will be carried out in pretrial detention facilities in the cantons of Zurich and Bern and aims to improve the wellbeing and social integration of individuals in pretrial detention. As part of the MV the investigators are evaluating the impact of two interventions using a randomized controlled trial (RCT). The first intervention, "Prison Stress Management" (PRISMA), addresses the issue of poor mental health of inmates during pretrial detention and after release. PRISMA is a scalable World Health Organization (WHO)-developed psychological intervention based on cognitive-behavioral therapy (CBT) program and goes beyond the status-quo mental health support offered in jails. Currently, only inmates with severe mental health problems are referred to the psychiatric ward of the health services provided in jails and no continuation of support is offered after the transition to the outside world. The second intervention (SOCIAL) uses extended social services to address potential disruptions incarceration might cause in detainees' social and economic lives. The isolation from the outside world implies that detainees might lose their jobs and housing, their relationships with their family and friends are strained, all factor hindering re-integration into society and taxing their mental wellbeing.

The present pilot RCT aims to investigate the feasibility and acceptability of an PRISMA for inmates to inform a full-scale, definitive randomized controlled trial. Data will be collected regarding the feasibility and acceptability of all study components, including recruitment, drop-out rate, protocol adherence, study visit attendance and the time burden of parent questionnaires. These data will inform the design of a full scale randomized controlled trial to evaluate the efficacy of PRISMA in inmates.

For this purpose only 20 people in each arm will be included.

ELIGIBILITY:
Inclusion Criteria:

* Entering pretrial detention inmate in any of the 11 pretrial detention facilities in the Cantons of Zurich and Bern
* aged ≥ 18 years

Exclusion Criteria:

* Not fluently speaking any of the nine languages in which PRISMA is offered: German, Albanian, Arabic, English, French, Italian, Romanian, Serbian/ Croatian, Spanish
* Acute suicidality
* Not interested in PRISMA and its randomized evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Verification procedure to the measurement in psychological distress | Three weeks (primary outcome) after intake; 10 weeks, and 6 months
  The primary outcome is mental health at three weeks as assessed by the scale for depression measured by Patient Health Questionnaire - 9 (PHQ9). A higher score on the PHQ9 (range = 1 - 27) means a greater severity of depressive symptoms.
Verification procedure to the measurement in psychological distress | Three weeks (primary outcome) after intake; 10 weeks, and 6 months
  The primary outcome is mental health at three weeks as assessed by the scale for anxiety, measured by Generalized Anxiety Disorder-7 (GAD-7). A higher score on the GAD-7 (range = 0 - 21) means a greater severity of anxiety symptoms.

SECONDARY OUTCOMES:
Verification procedure to the measurement suicidal ideation | Screening, 3 weeks follow-up assessment, 10 weeks, 6 months and 1 year after the intervention
  Suicidal Ideation is measured using an adapted version of the Suicidal Ideation Attribution Scale (SIDAS), a brief measure of severity of suicidal ideation assessing frequency, controllability, closeness to attempt, level of distress associated with the thoughts and impact on daily functioning. It consists of 3 items rated on an 11-point scale (0 = "Never" to 10 = "Always").
Feasibility of PRISMA by the number of dropouts | Screening, 3 weeks follow-up assessment, 10 weeks, 6 months and 1 year after the intervention
  Monitoring of the dropouts by number of participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided